CLINICAL TRIAL: NCT01710488
Title: A Randomized, Controlled, Single-blind, Parallel-group Comparison Between Levofloxacin and Prulifloxacin, in Patients With Acute Exacerbation of COPD Unresponsive to Other Antibiotics and Admitted to the Internal Medicine
Brief Title: Comparison Between Levofloxacin and Prulifloxacin, in Internal Medicine Patients With Acute Exacerbation of COPD
Acronym: FLOR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fadoi Foundation, Italy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EudraCT N. 2008-003842-27
Record Dates: First submitted 2012-10-12; First posted 2012-10-19 (Estimated); Results first posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2012-10

CONDITIONS: COPD Exacerbation
Keywords: COPD exacerbation; fluoroquinolones,

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levofloxacin 1 tablet 500 mg once a day (Active Comparator): Levofloxacin 1 tablet 500 mg once a day for 7-10 days. It will be used, according to a randomization list pre-ordered, centralized, in blocks of 4 patients
  Interventions: Drug: Levofloxacin 1 tablet 500 mg once a day
- Prulifloxacin 1 tablet 600 mg once a day (Experimental): Prulifloxacin 1 tablet 600 mg once a day for 7-10 days. It will be used, according to a randomization list pre-ordered, centralized, in blocks of 4 patients
  Interventions: Drug: Prulifloxacin 1 tablet 600 mg once a day

INTERVENTIONS:
Drug: Levofloxacin 1 tablet 500 mg once a day — Will be used, according to a randomization list pre-ordered, centralized, in blocks of 4 patients:
  Levofloxacin 500 mg (1 tablet) once daily for 7-10 days. The prescribing and dispensing of the drug will be made by medical personnel not directly involved in the data collection procedures for the study, and nursing staff, and the Medical Investigator will not be aware of the type of treatment to the individual. The drugs will be administered in the morning, about two hours after food.
  Other Names: LEVOXACIN 500 mg
  Arms: Levofloxacin 1 tablet 500 mg once a day
Drug: Prulifloxacin 1 tablet 600 mg once a day — Will be used, according to a randomization list pre-ordered, centralized, in blocks of 4 patients:
  Prulifloxacin 1 tablet 600 mg once daily for 7-10 days. The prescribing and dispensing of the drug will be made by medical personnel not directly involved in the data collection procedures for the study, and nursing staff, and the Medical Investigator will not be aware of the type of treatment to the individual. The drugs will be administered in the morning, about two hours after food.
  Other Names: UNIDROX 600 mg
  Arms: Prulifloxacin 1 tablet 600 mg once a day

SUMMARY:
The primary objective of the study is to determine the percentage of patients with "therapeutic success" at the end of the cycle of antibiotic therapy (10 days), in the two treatment groups (levofloxacin and prulifloxacin). The effect of study treatments will be evaluated on the basis of a score determined in relation to the signs-symptoms of acute exacerbation of COPD (sputum purulence, sputum volume, cough, dyspnea, fever)

DETAILED DESCRIPTION:
The aim of this study was to examine the effects of the use of fluoroquinolones a class of antibiotics introduced relatively recently, in a particular population of patients with acute exacerbation of COPD, previously treated unsuccessfully with other antibiotics, and hospitalized in Internal Medicine. These patients reflect the reality of patients admitted to Internal Medicine, they are characterized by a high frequency of advanced age, polypathology, with multiple treatments.

ELIGIBILITY:
Inclusion Criteria:

* - Presence of purulent sputum documented by colorimetric assay (Allegra et al., Resp Med 2005), plus at least two of the following signs-symptoms
* Increased cough
* Increased dyspnea
* Increase in sputum volume appeared at least 3 days
* previous antibiotic treatment with any medication (eg, amoxicillin, amoxicillin / clavulanate, cephalosporins or macrolides) with the exception of quinolones, conducted for at least 3 days with persistence or worsening of symptoms and subsequent use of hospital
* ≥ 60 years
* FEV1 <80% and ≥ 30% and ratio FEV 1 / FVC <70%
* chest x-ray negative for inflammatory infiltrates
* informed consent

Exclusion Criteria:

* asthma
* pulmonary neoplasms
* a history of allergy or hypersensitivity to quinolones
* impracticability in oral antibiotic and / or altered ability to absorption by the gastrointestinal system
* a history of epilepsy, seizures, cerebral vascular disease (stroke cerebri within 6 months)
* history of tendinopathy
* note or severe renal impairment creatinine> than twice the upper limit of the normal range or hepatic impairment (AST and / or ALT> twice the upper limit of the normal range)
* patients with sepsis, tuberculosis or other infections in other organs or systems
* cystic fibrosis
* patients with inherited tolerance to intolerance, Lapp lactase deficiency or glucose-galactose malabsorption, or deficiency of the enzyme glucose-6-phosphate dehydrogenase
* pregnant or breastfeeding
* drug or alcohol addiction
* experimental concomitant treatment with other drugs

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2009-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gualberto GG Gussoni, MD, PhD, Study Director — Dept. Clinical Research "Study Centre" - FadoiFoundation
Locations (25):
- Italy (25):
  - Hospita "San Francesco Caracciolo", Agnone
  - Hospital of Alghero, Alghero
  - Hospital "Cardinal Massaia", Asti
  - Hospital "Fatebenefratelli", Benevento
  - Hospital of Bordighera, Bordighera
  - Hospital "San Giovanni di Dio", Cagliari
  - Hospital "Pugliese-Ciaccio", Catanzaro
  - Hospital "L.Parodi Delfino", Colleferro
  - Hospita "San Giovanni di Dio", Crotone
  - Hospital "E.Profili" of Fabriano, Fabriano
  - Hospital "F. Veneziale", Isernia
  - Hospital Civile Legnano, Legnano
  - Hospital of Ortona, Ortona
  - Hospital Fatebenefratelli "Buccheri La Ferla", Palermo
  - Hospital "Sant'Anna", Reggio Emilia
  - Hospital " Santa Maria Nuova", Reggio Emilia
  - Hospital "Policlinico Universitario Campus Biomedico", Rome
  - Hospital "Casa Sollievo della Sofferenza", San Giovanni Rotondo
  - Hospital of Scandiano, Scandiano
  - Hospital "Paolo Dettori", Tempio Pausania
  - Hospital "Santa Maria" of Terni, Terni
  - Hospital "San Giovanni Bosco", Torino
  - Hospital "Jazzolino", Vibo Valentia
  - Hospital "San Bortolo", Vicenza
  - Hospital "Santa Maria Maddalena", Volterra

RESULTS

PARTICIPANT FLOW:
Groups:
- Levofloxacin 1 Tablet 500 mg Once a Day: Levofloxacin 1 tablet 500 mg once a day for 7-10 days. It will be used, according to a randomization list pre-ordered, centralized, in blocks of 4 patients
  Levofloxacin 1 tablet 500 mg once a day: Will be used, according to a randomization list pre-ordered, centralized, in blocks of 4 patients:
  Levofloxacin 500 mg (1 tablet) once daily for 7-10 days. The prescribing and dispensing of the drug will be made by medical personnel not directly involved in the data collection procedures for the study, and nursing staff, and the Medical Investigator will not be aware of the type of treatment to the individual. The drugs will be administered in the morning, about two hours after food.
- Prulifloxacin 1 Tablet 600 mg Once a Day: Prulifloxacin 1 tablet 600 mg once a day for 7-10 days. It will be used, according to a randomization list pre-ordered, centralized, in blocks of 4 patients
  Prulifloxacin 1 tablet 600 mg once a day: Will be used, according to a randomization list pre-ordered, centralized, in blocks of 4 patients:
  Prulifloxacin 1 tablet 600 mg once daily for 7-10 days. The prescribing and dispensing of the drug will be made by medical personnel not directly involved in the data collection procedures for the study, and nursing staff, and the Medical Investigator will not be aware of the type of treatment to the individual. The drugs will be administered in the morning, about two hours after food.
Period: Overall Study
Arm/Group | Levofloxacin 1 Tablet 500 mg Once a Day | Prulifloxacin 1 Tablet 600 mg Once a Day
Started | 128 | 130
Completed | 92 | 96
Not Completed | 36 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levofloxacin 1 Tablet 500 mg Once a Day | Prulifloxacin 1 Tablet 600 mg Once a Day | Total
Number analyzed (Participants) | 128 | 130 | 258
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 119 | 121 | 240
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 39 | 76
  Male | 91 | 91 | 182
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Italy | 128 | 130 | 258

OUTCOME MEASURES:

1. Primary Outcome: The Primary Objective of the Study is to Determine the Percentage of Patients With "Therapeutic Success" at the End of the Cycle of Antibiotic Therapy (10 Days), in the Two Treatment Groups (Levofloxacin and Prulifloxacin).
Description: The effect of study treatments will be evaluated on the basis of a score determined in relation to the signs-symptoms of acute exacerbation of COPD (sputum purulence, sputum volume, cough, dyspnea, fever). The primary study end-point was the percentage of patients with "therapeutic success" (disappearance of all signs/symptoms of disease or reduction of at least 3 points of the total score of symptomatology from baseline) at the conclusion of the cycle of antibiotic therapy (day 10), in the two study groups (levofloxacin and prulifloxacin).
Time Frame: 10 days
Population: The analyses concerning the primary study end-point were carried out both on the "intention-to-treat" and "per-protocol" populations, more than 90% of patients had a therapeutic success at the end of treatment cycle in both study groups. Here is reported the ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Levofloxacin 1 Tablet 500 mg Once a Day | Prulifloxacin 1 Tablet 600 mg Once a Day
Number analyzed (Participants) | 128 | 130
Participants | 119 | 126

2. Secondary Outcome: Percentage of Successful Treatment to Day 7 of Treatment
Time Frame: 7 days
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Rehospitalization for COPD Exacerbation During the Follow-up
Time Frame: one year
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Number of Episodes of Exacerbations
Time Frame: one year
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Additional Cycles of Antibiotic
Time Frame: one year
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Survival
Time Frame: one year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Total time frame for adeverse drug reaction: 10 days or 7 days + 1 month Total time frame for survival: 10 days or 7 days + 1 year
Description: Adverse event and/or serious adverse event, used to collect adverse event information, not differs from the clinicaltrials.gov
Arm/Group | Levofloxacin 1 Tablet 500 mg Once a Day | Prulifloxacin 1 Tablet 600 mg Once a Day
All-Cause Mortality (participants affected / at risk) | 11/128 | 5/130
Serious Adverse Events (participants affected / at risk) | 2/128 | 1/130
Other Adverse Events (participants affected / at risk) | 1/128 | 5/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levofloxacin 1 Tablet 500 mg Once a Day (N=128) | Prulifloxacin 1 Tablet 600 mg Once a Day (N=130)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Acute renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levofloxacin 1 Tablet 500 mg Once a Day (N=128) | Prulifloxacin 1 Tablet 600 mg Once a Day (N=130)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Psychomotor agitation (Nervous system disorders) | 0 (0) | 1 (1)
muscular pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Epigastric pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No